CLINICAL TRIAL: NCT04551001
Title: Randomized Controlled Trial Investigating Cold Snare aNd Forcep polypectomY Among Small POLYPs in Rates of Complete Resection: the TINYPOLYP Trial.
Brief Title: Evaluation of Cold Forcep and Cold Snare Polypectomy for Polyps Less Than or Equal to 3mm in Size During Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Shai Friedland, Professor in Gastroenterology & Hepatology, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15766-1
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Colo-rectal Cancer; Polyp of Colon; Adenomatous Polyp of Colon
MeSH Terms: conditions — Colonic Neoplasms; Colonic Polyps

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cold forcep (Experimental): Cold forcep polypectomy performed for polyps <=3mm.
  Interventions: Procedure: Cold forcep polypectomy
- Cold snare (Experimental): Cold forcep polypectomy performed for polyps <=3mm.
  Interventions: Procedure: Cold snare polypectomy

INTERVENTIONS:
Procedure: Cold forcep polypectomy — Removal of appropriate polyps using cold forceps until no polyp visible under white light. Two additional biopsies performed at margins of polypectomy site.
  Arms: Cold forcep
Procedure: Cold snare polypectomy — Removal of appropriate polyps using cold snare until no polyp visible under white light. Two additional biopsies performed at margins of polypectomy site.
  Arms: Cold snare

SUMMARY:
The focus of the study is to evaluate impact of cold forcep and cold snare in achieving complete resection during polypectomy of polyps <=3mm during colonoscopy.

DETAILED DESCRIPTION:
The details of the proposed study are as follows:

1. Experimental group: using cold forceps for polyps <=3mm of the colon
2. Control group: using cold snare for polyps <=3mm of the colon
3. Methods:

   1. Colonoscopy will be performed in the same standard of care manner as if no study was taking place.
   2. If polyps <=3mm are identified, the endoscopist is randomized to performing polypectomy with cold forcep or cold snare.
   3. After removal of the polypectomy, two biopsies are performed at the margin of the polypectomy site to identify residual lesion.
   4. The polyp as well as well as the two biopsies are reviewed by a pathologist.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older
* Polyps <=3mm

Exclusion Criteria:

* Pregnant
* Inflammatory bowel disease
* Polyposis syndromes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-11-20 (Actual)

PRIMARY OUTCOMES:
Completeness of resection | 2 weeks
  The primary outcome measured is comparison of completeness of resection between the cold forcep and cold snare groups.

SECONDARY OUTCOMES:
Time to resection | During the procedure
  The time between the forceps or snare is introduced till the polyp is removed and retrieved will be compared.
Number of forcep bites or snare attempts | During the procedure
  We will compare the number of bites or snare attempts needed to remove the tissue adequately to the endoscopist's judgment.
Complications | 4 weeks
  We will compare rates of complications including perforation and immediate post-polypectomy bleeding, early post-polypectomy bleed (within 24 hours) and delayed post polypectomy bleed (between 24 hours and 30 days). Early post-polypectomy bleed and delayed post-polypectomy bleed is evaluated based on emergency room (ER) visit, inpatient stay, transfusion needed, repeat colonoscopy required, surgical intervention required, and mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Shai Friedland, MD, Principal Investigator — Stanford University
Locations (1):
- Veterans Affairs Palo Alto Health Care System, Palo Alto, California, United States

REFERENCES:
- [Derived] Wei MT, Louie CY, Chen Y, Pan JY, Quan SY, Wong R, Brown R, Clark M, Jensen K, Lau H, Friedland S. Randomized Controlled Trial Investigating Cold Snare and Forceps Polypectomy Among Small POLYPs in Rates of Complete Resection: The TINYPOLYP Trial. Am J Gastroenterol. 2022 Aug 1;117(8):1305-1310. doi: 10.14309/ajg.0000000000001799. Epub 2022 Apr 25. PMID 35467557